CLINICAL TRIAL: NCT02549755
Title: Feasibility of 11C-acetate in the Monitoring of Treatment Response Following Radiotherapy in Patients With Hepatocellular Carcinoma
Brief Title: 11C-acetate for Treatment Response After Radiotherapy for HCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Justin Sims (Other)
Responsible Party: Sponsor-Investigator, Justin Sims, Assistant Professor of Clinical Radiology, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IUSCC-0543
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — carbon-11 acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy treatment monitoring of hepatocellular carcinoma (Other): All patients enrolled in the trial will undergo 3 PET/CT studies using 11C-acetate at the injected radiotracer. The patients will be imaged prior to their radiation therapy and at 1 and 3 months following the completion of their radiation therapy. They will also undergo an MRI scan of the liver at each of those time points.
  Interventions: Drug: 11C-Acetate

INTERVENTIONS:
Drug: 11C-Acetate — The 11C-Acetate radiopharmaceutical will be administered intravenously at a dose of 20-40 mCi (0.74-1.5 GBq).
  There will be a total of three 11C-acetate radiopharmaceutical administrations for each patient

SUMMARY:
It is thought that PET of the abdomen with 11C Acetate will provide new information regarding whether or not patient's have benefited from radiotherapy. To test this theory, the project will evaluate the potential of 11C acetate to serve as an earlier and/or better signal of treatment success.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Subject is willing to participate in the study and has signed the study informed consent
* Subject is available and willing to comply with the protocol evaluations
* Diagnosed hepatocellular carcinoma confined to a single lobe of the liver if undergoing 90Y radioembolization
* Diagnosed hepatocellular carcinoma confined to the liver if undergoing Stereotactic Body Radiation Therapy (SBRT)
* Under consideration for 90Y radioembolization or Stereotactic Body Radiation Therapy (SBRT)

Exclusion Criteria:

* Pregnant or planning to become pregnant within the next 12 months or breast-feeding
* GFR < 45
* Life expectancy < 6 months
* Claustrophobic and cannot tolerate imaging procedures
* Weigh > 350 lb (upper weight limit of scanner beds)
* Special vulnerabilities (e.g. fetuses, neonatales, pregnant women, children, prisoners, institutionalized individuals).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin B Sims, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Dancey JE, Shepherd FA, Paul K, Sniderman KW, Houle S, Gabrys J, Hendler AL, Goin JE. Treatment of nonresectable hepatocellular carcinoma with intrahepatic 90Y-microspheres. J Nucl Med. 2000 Oct;41(10):1673-81. PMID 11037997
- [Background] Andolino DL, Johnson CS, Maluccio M, Kwo P, Tector AJ, Zook J, Johnstone PA, Cardenes HR. Stereotactic body radiotherapy for primary hepatocellular carcinoma. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e447-53. doi: 10.1016/j.ijrobp.2011.04.011. Epub 2011 Jun 7. PMID 21645977
- [Background] Forner A, Ayuso C, Varela M, Rimola J, Hessheimer AJ, de Lope CR, Reig M, Bianchi L, Llovet JM, Bruix J. Evaluation of tumor response after locoregional therapies in hepatocellular carcinoma: are response evaluation criteria in solid tumors reliable? Cancer. 2009 Feb 1;115(3):616-23. doi: 10.1002/cncr.24050. PMID 19117042
- [Background] Llovet JM, Di Bisceglie AM, Bruix J, Kramer BS, Lencioni R, Zhu AX, Sherman M, Schwartz M, Lotze M, Talwalkar J, Gores GJ; Panel of Experts in HCC-Design Clinical Trials. Design and endpoints of clinical trials in hepatocellular carcinoma. J Natl Cancer Inst. 2008 May 21;100(10):698-711. doi: 10.1093/jnci/djn134. Epub 2008 May 13. PMID 18477802
- [Background] Riaz A, Miller FH, Kulik LM, Nikolaidis P, Yaghmai V, Lewandowski RJ, Mulcahy MF, Ryu RK, Sato KT, Gupta R, Wang E, Baker T, Abecassis M, Benson AB 3rd, Nemcek AA Jr, Omary R, Salem R. Imaging response in the primary index lesion and clinical outcomes following transarterial locoregional therapy for hepatocellular carcinoma. JAMA. 2010 Mar 17;303(11):1062-9. doi: 10.1001/jama.2010.262. PMID 20233824
- [Background] Keppke AL, Salem R, Reddy D, Huang J, Jin J, Larson AC, Miller FH. Imaging of hepatocellular carcinoma after treatment with yttrium-90 microspheres. AJR Am J Roentgenol. 2007 Mar;188(3):768-75. doi: 10.2214/AJR.06.0706. PMID 17312067
- [Background] Krinsky GA, Lee VS, Theise ND, Weinreb JC, Rofsky NM, Diflo T, Teperman LW. Hepatocellular carcinoma and dysplastic nodules in patients with cirrhosis: prospective diagnosis with MR imaging and explantation correlation. Radiology. 2001 May;219(2):445-54. doi: 10.1148/radiology.219.2.r01ma40445. PMID 11323471
- [Background] Peterson MS, Baron RL, Marsh JW Jr, Oliver JH 3rd, Confer SR, Hunt LE. Pretransplantation surveillance for possible hepatocellular carcinoma in patients with cirrhosis: epidemiology and CT-based tumor detection rate in 430 cases with surgical pathologic correlation. Radiology. 2000 Dec;217(3):743-9. doi: 10.1148/radiology.217.3.r00dc28743. PMID 11110938
- [Background] Fendler WP, Philippe Tiega DB, Ilhan H, Paprottka PM, Heinemann V, Jakobs TF, Bartenstein P, Hacker M, Haug AR. Validation of several SUV-based parameters derived from 18F-FDG PET for prediction of survival after SIRT of hepatic metastases from colorectal cancer. J Nucl Med. 2013 Aug;54(8):1202-8. doi: 10.2967/jnumed.112.116426. Epub 2013 May 31. PMID 23729697
- [Background] Verhoef C, Valkema R, de Man RA, Krenning EP, Yzermans JN. Fluorine-18 FDG imaging in hepatocellular carcinoma using positron coincidence detection and single photon emission computed tomography. Liver. 2002 Feb;22(1):51-6. doi: 10.1046/j.0106-9543.2001.01593.x. PMID 11906619
- [Background] Khan MA, Combs CS, Brunt EM, Lowe VJ, Wolverson MK, Solomon H, Collins BT, Di Bisceglie AM. Positron emission tomography scanning in the evaluation of hepatocellular carcinoma. J Hepatol. 2000 May;32(5):792-7. doi: 10.1016/s0168-8278(00)80248-2. PMID 10845666
- [Background] Trojan J, Schroeder O, Raedle J, Baum RP, Herrmann G, Jacobi V, Zeuzem S. Fluorine-18 FDG positron emission tomography for imaging of hepatocellular carcinoma. Am J Gastroenterol. 1999 Nov;94(11):3314-9. doi: 10.1111/j.1572-0241.1999.01544.x. PMID 10566736
- [Background] Larsson P, Arvidsson D, Bjornstedt M, Isaksson B, Jersenius U, Motarjemi H, Jacobsson H. Adding 11C-acetate to 18F-FDG at PET Examination Has an Incremental Value in the Diagnosis of Hepatocellular Carcinoma. Mol Imaging Radionucl Ther. 2012 Apr;21(1):6-12. doi: 10.4274/Mirt.87. Epub 2012 Apr 1. PMID 23487415
- [Background] Ho CL, Yu SC, Yeung DW. 11C-acetate PET imaging in hepatocellular carcinoma and other liver masses. J Nucl Med. 2003 Feb;44(2):213-21. PMID 12571212
- [Background] Ho CL, Chen S, Yeung DW, Cheng TK. Dual-tracer PET/CT imaging in evaluation of metastatic hepatocellular carcinoma. J Nucl Med. 2007 Jun;48(6):902-9. doi: 10.2967/jnumed.106.036673. Epub 2007 May 15. PMID 17504862
- [Background] Park JW, Kim JH, Kim SK, Kang KW, Park KW, Choi JI, Lee WJ, Kim CM, Nam BH. A prospective evaluation of 18F-FDG and 11C-acetate PET/CT for detection of primary and metastatic hepatocellular carcinoma. J Nucl Med. 2008 Dec;49(12):1912-21. doi: 10.2967/jnumed.108.055087. Epub 2008 Nov 7. PMID 18997056
- [Background] Cheung TT, Ho CL, Lo CM, Chen S, Chan SC, Chok KS, Fung JY, Yan Chan AC, Sharr W, Yau T, Poon RT, Fan ST. 11C-acetate and 18F-FDG PET/CT for clinical staging and selection of patients with hepatocellular carcinoma for liver transplantation on the basis of Milan criteria: surgeon's perspective. J Nucl Med. 2013 Feb;54(2):192-200. doi: 10.2967/jnumed.112.107516. Epub 2013 Jan 15. PMID 23321459
- [Background] Mock BH, Brown-Proctor C, Green MA, Steele B, Glick-Wilson BE, Zheng QH. An automated SPE-based high-yield synthesis of [11C]acetate and [11C]palmitate: no liquid-liquid extraction, solvent evaporation or distillation required. Nucl Med Biol. 2011 Nov;38(8):1135-42. doi: 10.1016/j.nucmedbio.2011.05.007. Epub 2011 Aug 9. PMID 21831651
- [Background] Tollinger CD, Vreman HJ, Weiner MW. Measurement of acetate in human blood by gas chromatography: effects of sample preparation, feeding, and various diseases. Clin Chem. 1979 Oct;25(10):1787-90. PMID 476928
- [Background] Jadvar H, Alavi A. Role of Imaging in Prostate Cancer. PET Clin. 2009 Apr 1;4(2):135-8. doi: 10.1016/j.cpet.2009.05.003. No abstract available. PMID 20161047
- [Background] Engelbrecht MR, Barentsz JO, Jager GJ, van der Graaf M, Heerschap A, Sedelaar JP, Aarnink RG, de la Rosette JJ. Prostate cancer staging using imaging. BJU Int. 2000 Jul;86 Suppl 1:123-34. doi: 10.1046/j.1464-410x.2000.00592.x. No abstract available. PMID 10961282
- [Background] Jadvar H. Prostate cancer: PET with 18F-FDG, 18F- or 11C-acetate, and 18F- or 11C-choline. J Nucl Med. 2011 Jan;52(1):81-9. doi: 10.2967/jnumed.110.077941. Epub 2010 Dec 13. PMID 21149473
- [Background] Oyama N, Miller TR, Dehdashti F, Siegel BA, Fischer KC, Michalski JM, Kibel AS, Andriole GL, Picus J, Welch MJ. 11C-acetate PET imaging of prostate cancer: detection of recurrent disease at PSA relapse. J Nucl Med. 2003 Apr;44(4):549-55. PMID 12679398
- [Background] Sandblom G, Sorensen J, Lundin N, Haggman M, Malmstrom PU. Positron emission tomography with C11-acetate for tumor detection and localization in patients with prostate-specific antigen relapse after radical prostatectomy. Urology. 2006 May;67(5):996-1000. doi: 10.1016/j.urology.2005.11.044. PMID 16698359
- [Background] Seltzer MA, Jahan SA, Sparks R, Stout DB, Satyamurthy N, Dahlbom M, Phelps ME, Barrio JR. Radiation dose estimates in humans for (11)C-acetate whole-body PET. J Nucl Med. 2004 Jul;45(7):1233-6. PMID 15235071
- [Background] Walsh MN, Geltman EM, Brown MA, Henes CG, Weinheimer CJ, Sobel BE, Bergmann SR. Noninvasive estimation of regional myocardial oxygen consumption by positron emission tomography with carbon-11 acetate in patients with myocardial infarction. J Nucl Med. 1989 Nov;30(11):1798-808. PMID 2809744
- [Background] Wang CL, Cohan RH, Ellis JH, Adusumilli S, Dunnick NR. Frequency, management, and outcome of extravasation of nonionic iodinated contrast medium in 69,657 intravenous injections. Radiology. 2007 Apr;243(1):80-7. doi: 10.1148/radiol.2431060554. PMID 17392249

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Arm: Enrolled patients are to undergo 3 acetate PET/CT examinations--the first within one month prior to radiotherapy, the second one month following, and the third three months following radiotherapy.
Period: Overall Study
Arm/Group | Main Arm
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: 1 adult male (greater than 18 years) meeting inclusion/exclusion criteria
Groups:
- Radiotherapy Treatment Monitoring of Hepatocellular Carcinoma: All patients enrolled in the trial will undergo 3 PET/CT studies using 11C-acetate at the injected radiotracer. The patients will be imaged prior to their radiation therapy and at 1 and 3 months following the completion of their radiation therapy. They will also undergo an MRI scan of the liver at each of those time points.
  11C-Acetate: The 11C-Acetate radiopharmaceutical will be administered intravenously at a dose of 20-40 mCi (0.74-1.5 GBq).
  There will be a total of three 11C-acetate radiopharmaceutical administrations for each patient
Arm/Group | Radiotherapy Treatment Monitoring of Hepatocellular Carcinoma
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1
Number of participants [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: To Compare Changes in 11C-acetate Uptake at One and Three Months Following Radiotherapy With Pre-treatment Uptake of 11C-acetate
Description: The single patient enrolled in the trial showed no uptake in the liver tumor on the pretreatment scan and was dropped from the trial.
Time Frame: At three months
Groups:
- Main Arm: The single patient enrolled in the trial did not show tumor uptake on the initial scan and was thus dropped from the trial. The study was terminated in November of 2016.
Arm/Group | Main Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the period of observation of the participant immediately before, during, and after the single PET/CT scan.
Groups:
- Main Arm: No adverse events occurred during the trial.
Arm/Group | Main Arm
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes